CLINICAL TRIAL: NCT00837512
Title: Insulin Delivery Using Microneedles in Type 1 Diabetes
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Eric Felner, MD, MSCR, Pediatric Endocrinology, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1348-2005; FWA00005792 (Other: Other)
Record Dates: First submitted 2009-02-04; First posted 2009-02-05 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2013-11

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: microneedle continuous subcutaneous insulin infusion
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Microneedle (Experimental): Microneedle used to deliver insulin at a depth less than 900 micrometers
  Interventions: Device: Microneedle
- Subcutaneous insulin catheter (Active Comparator): Subcutaneous insulin catheter used to deliver insulin at a depth of 9 mm (9000 micrometers)
  Interventions: Device: Subcutaneous insulin catheter

INTERVENTIONS:
Device: Microneedle — Microneedle used to deliver insulin at a depth less than 900 micrometers
  Arms: Microneedle
Device: Subcutaneous insulin catheter — Subcutaneous insulin catheter used to deliver insulin at a depth of 9 mm (9000 micrometers)
  Other Names: subcutaneous insulin infusion catheter
  Arms: Subcutaneous insulin catheter

SUMMARY:
The goal of this study is to determine if microneedles can effectively and painlessly deliver insulin to children and young adults with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 8 years of age
* <19 years of age
* Type 1 Diabetes for at least 2 years
* Uses a conventional, FDA-approved insulin pump for the past year
* Uses Lispro insulin
* Mean hemoglobin A1C ≤ 8.5 % for the past year
* Body mass index ≤ 85th percentile for age
* Understand and be willing to adhere to the study protocol

Exclusion Criteria:

* Type 2 Diabetes
* Acanthosis nigricans
* Clinically significant major organ system disease
* On glucocorticoid therapy
* Insulin requirement ≥ 150 U/day
* Illness on the day of the study
* Cognitive impairment (IQ < 85 or > 2 grades behind age-appropriate grade)
* Pregnant or breast-feeding (if female).

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2008-09; Primary Completion 2012-12 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Emory University, Atlanta, Georgia, United States

REFERENCES:
- [Derived] Norman JJ, Brown MR, Raviele NA, Prausnitz MR, Felner EI. Faster pharmacokinetics and increased patient acceptance of intradermal insulin delivery using a single hollow microneedle in children and adolescents with type 1 diabetes. Pediatr Diabetes. 2013 Sep;14(6):459-65. doi: 10.1111/pedi.12031. Epub 2013 Mar 21. PMID 23517449

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from our outpatient clinic setting within the Emory Children's Center
Pre-assignment Details: In the event that the potential subject was on Humalog they switched to Novolog 48 hours prior to first visit.
Groups:
- First: Microneedle: Microneedle : Microneedle used to deliver insulin at a depth less than 900 micrometers
- First: Subcutaneous Insulin Catheter: Subcutaneous insulin catheter : Subcutaneous insulin catheter used to deliver insulin at a depth of 9 mm (9000 micrometers)
Period: First Intervention (6hrs) - RANDOMIZED
Arm/Group | First: Microneedle | First: Subcutaneous Insulin Catheter
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: Both Arms: Washout (7-28 Days)
Arm/Group | First: Microneedle | First: Subcutaneous Insulin Catheter
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0
Period: 2nd Intervention (6 Hrs) - RANDOMIZED
Arm/Group | First: Microneedle | First: Subcutaneous Insulin Catheter
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Microneedle : Microneedle used to deliver insulin at a depth less than 900 micrometers Subcutaneous insulin catheter : Subcutaneous insulin catheter used to deliver insulin at a depth of 9 mm (9000 micrometers)
Arm/Group | Entire Study Population
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.61 (2.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 16
Microneedle [Number; unit: Participants] — Subcutaneous insulin catheter used to deliver insulin at a depth of 9 mm (9000 micrometers)
  Participants
    Female | 7
    Male | 9
Subcutaneous insulin catheter [Number; unit: participants] — Subcutaneous insulin catheter used to deliver insulin at a depth of 9 mm (9000 micrometers)
  participants
    Female | 7
    Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Onset Time (Tmax)
Description: Average time to peak insulin concentration
Time Frame: 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 2.5, 3, 3.5, 4 hours
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Microneedle: Microneedle : Microneedle used to deliver insulin at a depth less than 900 micrometers
- Subcutaneous Insulin Catheter: Subcutaneous insulin catheter : Subcutaneous insulin catheter used to deliver insulin at a depth of 9 mm (9000 micrometers)
Arm/Group | Microneedle | Subcutaneous Insulin Catheter
Number analyzed (Participants) | 12 | 12
Minutes | 30 (2) | 52 (4)

ADVERSE EVENTS:
Arm/Group | Microneedle | Subcutaneous Insulin Catheter
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No